CLINICAL TRIAL: NCT01825356
Title: Amniotic Membrane as an Adjunct Treatment for Hallux Rigidus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-13-03A
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dorsal Cheilectomy no Amniotic Membrane Tissue Implantation (Active Comparator): Dorsal cheilectomy is a surgery for hallux rigidus(degenerative arthritis and stiffness due to bone spurs that affect the joint at the base of the big toe). No amniotic membrane will be used for this group.
  Interventions: Procedure: Dorsal Cheilectomy without Amniotic Membrane Tissue Implantation
- Dorsal Cheilectomy-Amniotic Membrane Tissue Implantation (Experimental): Dorsal cheilectomy procedure with the addition of the amniotic membrane. Amniotic membrane represents a biologic therapy that has the ability to actively regulate myrofibroblast formation and activity within the joint space and surgical site
  Interventions: Procedure: Dorsal Cheilectomy with Amniotic Membrane Tissue Implantation

INTERVENTIONS:
Procedure: Dorsal Cheilectomy without Amniotic Membrane Tissue Implantation
  Arms: Dorsal Cheilectomy no Amniotic Membrane Tissue Implantation
Procedure: Dorsal Cheilectomy with Amniotic Membrane Tissue Implantation
  Arms: Dorsal Cheilectomy-Amniotic Membrane Tissue Implantation

SUMMARY:
The purpose of this study is to determine whether patients undergoing a dorsal cheilectomy procedure with implementation of amniotic membrane tissue results in improved clinical and functional outcomes compared to a standard dorsal cheilectomy procedure.

Specific Aim 1:

To compare American Orthopedic Foot and Ankle Society (AOFAS) scores between patients undergoing dorsal cheilectomy to patients undergoing dorsal cheilectomy with implantation of amniotic membrane tissue.

Hypothesis 1: Clinical and functional outcomes, as measured by the AOFAS , in the patients undergoing dorsal cheilectomy with implantation of amniotic membrane tissue will be superior to those without.

Specific Aim 2:

To compare range of motion between patients undergoing dorsal cheilectomy to patients undergoing dorsal cheilectomy with implantation of amniotic membrane tissue.

Hypothesis 2: Patient to undergo dorsal cheilectomy and implantation of amniotic membrane tissue will demonstrate less postoperative stiffness as measured from the pre-and postoperative radiographs.

Specific Aim 3:

To compare Foot Function Index (FFI) scores between patients undergoing dorsal cheilectomy to patients undergoing dorsal cheilectomy with implantation of amniotic membrane tissue.

Hypothesis 3: Clinical and functional outcomes, as measured by the FFI, the patients undergoing dorsal cheilectomy with implantation of amniotic membrane tissue will be superior to those without.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with an isolated diagnosis of type II hallux rigidus who are candidates for operative management with dorsal cheilectomy.
* Patients over the age of 18 able to consent to participate
* The subject is psychosocially, mentally, and physically able to understand and comply with the requirements of the study

Exclusion Criteria:

* < 18 years of age
* Patients that use ambulatory assistive devices
* Patients with systemic inflammtory arthritis
* Patient undergoing revision surgery for hallux rigidus to the ipsilateral extremity
* Patients with significant arthritis requiring alternative surgery other than dorsal cheilectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) score | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: John K Ellington, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States